CLINICAL TRIAL: NCT03751007
Title: A Prospective, Multi-center, Phase 1b/2a Study to Assess the Safety and Tolerability of Different Doses of AG019 Administered Alone or in Association With Teplizumab in Patients With Clinical Recent-onset Type 1 Diabetes Mellitus (T1D)
Brief Title: A Study to Assess the Safety and Tolerability of Different Doses of AG019 Administered Alone or in Combination With Teplizumab in Participants With Recent-onset Diagnosed Type 1 Diabetes (T1D)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Precigen Actobio T1D, LLC (Industry)
Collaborators: Intrexon Actobiotics NV, d/b/a Precigen Actobio (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG019-T1D-101; 2017-002871-24 (EudraCT Number)
Record Dates: First submitted 2018-11-08; First posted 2018-11-23 (Actual); Results first posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Diabetes type1
MeSH Terms: interventions — teplizumab

STUDY DESIGN:
Intervention Model Description: The phase 1b part of the study will enroll 4 sequential AG019 cohorts of up to 6 participants, in ascending dose cohorts and descending age cohorts. All participants in these cohorts will be treated with AG019 in an open label fashion.
  The phase 2a part of the study will evaluate 2 cohorts of participants administered AG019 and teplizumab. The first 2 participants will be treated with active treatment in an open label fashion. Participants 3-12 will be randomized (4:1) to receive active treatment or placebo in a double-blind fashion.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: For the randomized participants in the combination cohorts, blinding will be accomplished by arranging for AG019 and placebo components as well as teplizumab and placebo components to have identical packaging.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- AG019 Cohort 1 - Low Dose/Adults (Experimental)
  Interventions: Biological: AG019 - Low Dose
- AG019 Cohort 2 - High Dose/Adults (Experimental)
  Interventions: Biological: AG019 - High Dose
- AG019 Cohort 3 - Low Dose/Adolescents (Experimental)
  Interventions: Biological: AG019 - Low Dose
- AG019 Cohort 4 - High Dose/Adolescents (Experimental)
  Interventions: Biological: AG019 - High Dose
- Combination Cohort 1 - Adults (Experimental)
  Interventions: Drug: Teplizumab; Drug: Placebo-AG019; Drug: Placebo-Teplizumab; Biological: AG019 - High Dose
- Combination Cohort 2 - Adolescents (Experimental)
  Interventions: Drug: Teplizumab; Drug: Placebo-AG019; Drug: Placebo-Teplizumab; Biological: AG019 - High Dose

INTERVENTIONS:
Biological: AG019 - Low Dose — Solid, orally administered capsule - 2 capsules per day for 1 day (single dose) or 8 weeks (repeat dose)
  Arms: AG019 Cohort 1 - Low Dose/Adults; AG019 Cohort 3 - Low Dose/Adolescents
Drug: Teplizumab — Daily IV infusions of Teplizumab during the first 12 days of AG019 treatment. Total cumulative dose is approximately 17mg (dose calculation based on body surface area).
  Arms: Combination Cohort 1 - Adults; Combination Cohort 2 - Adolescents
Drug: Placebo-AG019 — Formulated identically to AG019 with the active ingredient removed.
  Arms: Combination Cohort 1 - Adults; Combination Cohort 2 - Adolescents
Drug: Placebo-Teplizumab — Formulated identically to teplizumab with the active ingredient removed.
  Arms: Combination Cohort 1 - Adults; Combination Cohort 2 - Adolescents
Biological: AG019 - High Dose — Solid, orally administered capsule - 6 capsules per day for 1 day (single dose) or 8 weeks
  Arms: AG019 Cohort 2 - High Dose/Adults; AG019 Cohort 4 - High Dose/Adolescents
Biological: AG019 - High Dose — Solid, orally administered capsule - 6 capsules per day for 8 weeks.
  Arms: Combination Cohort 1 - Adults; Combination Cohort 2 - Adolescents

SUMMARY:
The purpose of this study is to assess the safety and tolerability of different doses of AG019 administered alone or in combination with teplizumab in participants with recent-onset type 1 diabetes (T1D).

DETAILED DESCRIPTION:
This Phase 1b/2a, multi-center study will be conducted in participants with clinical recent-onset type 1 diabetes (T1D).

The primary objective of this study is to assess the safety and tolerability of different doses of AG019 alone as well as AG019 in combination with teplizumab. The secondary objectives of this study are: to obtain pharmacodynamic (PD) data of AG019 alone as well as AG019 in combination with teplizumab; and to determine the potential presence of AG019 in systemic circulation (safety - systemic exposure) and the presence of L. lactis bacteria in fecal excretion (local exposure): Pharmacokinetic (PK) profile.

This study consists of 2 phases:

Phase 1b: this open-label part of the study will investigate the safety and tolerability of 2 different doses of AG019 in 2 age groups (18-40 years of age and 12-17 years of age).

Phase 2a: this randomized, double-blind part of the study will investigate the safety and tolerability of AG019, in combination with teplizumab, in 2 age groups (18-40 years of age and 12-17 years of age).

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating females, 18 - 40 years of age (both inclusive) or 12-17 years of age (both inclusive)
* Diagnosis of diabetes according to the American Diabetes Association (ADA) recommended criteria
* Evidence of auto-antibodies to at least 1 β-cell autoantigen
* Stimulated C-peptide measured during 4h Mixed Meal tolerance Test (MMTT) > 0.2 nmol/L
* The first administration of AG019 should occur no later than 150 days post diagnosis of diabetes
* Body weight ≥ 33kg
* Written informed consent obtained and documented (participant, parent, guardian as applicable)

Exclusion Criteria:

* Previous history of serious cytokine release syndrome to teplizumab or other humanized anti-CD3 monoclonal antibodies with no or minimal capacity to bind Fc receptors. (Participants enrolled in the second phase of the trial in either Combination Cohort 1 or Combination Cohort 2, only)
* Use of immunosuppressive or immunomodulatory therapies, including systemic steroids within 1 month prior to randomization
* Participation in another investigational drug trial within 12 weeks prior to the first study drug intake and during participation in this study
* History of recurrent infections, other autoimmune diseases, cardiac disease, malignancy, or any other (chronic) medical condition which, in the investigator's opinion, could compromise participant safety
* Documented history of human immunodeficiency virus (HIV), Hepatitis Virus Type C (HCV), Hepatitis Virus Type B (HBV) infection
* Evidence of active infection with Epstein-Barr Virus (EBV) or cytomegalovirus (CMV)
* Evidence of active or latent tuberculosis (TB)
* Administration of anti-CD3 antibody in past year
* Current therapy with any other anti-diabetic agents other than insulin (MDI, CSII or analogue). Current or planned therapy with experimental (i.e., unapproved) insulin. Patients on therapy for type 2 diabetes (e.g. metformin) should stop their therapy in order to be eligible for study participation.
* Use of medications known to influence glucose tolerance
* Daily use of non-steroidal anti-inflammatory agents
* Compromised GI mucosal integrity or motility, not attributable to T1D (i.e., recent diarrhea, gluten sensitive enteropathy, inflammatory bowel disease, irritable bowel syndrome), or current use of medications known to influence GI motility
* Positive result of SARS-Cov2 PCR test at screening or within 3 days before randomization

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Mathieu, MD, Principal Investigator — University Hospital of Leuven, Clinical and Experimental Endocrinology; Kevan Herold, MD, Principal Investigator — Yale Center for Clinical Investigation; Yale University
Locations (18):
- United States (15):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - Coastal Metabolic Research Centre, Ventura, California
  - University of Colorado, Aurora, Colorado
  - Yale Center for Clinical Investigation, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Barry J Reiner, MD, LLC, Baltimore, Maryland
  - University of Minnesota Health, Minneapolis, Minnesota
  - University of Missouri-Kansas City School of Medicine, Kansas City, Missouri
  - Sanford Children's Specialty Clinic, Sioux Falls, South Dakota
  - University Diabetes and Endocrine Consultants, Chattanooga, Tennessee
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - Research Institute of Dallas, Dallas, Texas
  - Benaroya Research Institute, Seattle, Washington
- Belgium (3):
  - UZ Brussel, Brussels
  - UZ Antwerpen, Edegem
  - UZ Leuven, Leuven

REFERENCES:
- [Derived] Mathieu C, Wiedeman A, Cerosaletti K, Long SA, Serti E, Cooney L, Vermeiren J, Caluwaerts S, Van Huynegem K, Steidler L, Blomme S, Rottiers P, Nepom GT, Herold KC; AG019-T1D-101 Trial Investigators. A first-in-human, open-label Phase 1b and a randomised, double-blind Phase 2a clinical trial in recent-onset type 1 diabetes with AG019 as monotherapy and in combination with teplizumab. Diabetologia. 2024 Jan;67(1):27-41. doi: 10.1007/s00125-023-06014-2. Epub 2023 Oct 2. PMID 37782353
- [Derived] Alexander LM, van Pijkeren JP. Modes of therapeutic delivery in synthetic microbiology. Trends Microbiol. 2023 Feb;31(2):197-211. doi: 10.1016/j.tim.2022.09.003. Epub 2022 Oct 8. PMID 36220750

RESULTS

PARTICIPANT FLOW:
Recruitment Details: AG019 monotherapy cohorts: a total of 8 single dose patients and 19 repeat dose patients.
  AG019/teplizumab combination cohorts: a total of 18 patients
Pre-assignment Details: * 18-40y, or 12-17y
  * diagnosis of diabetes according to ADA criteria
  * positive for at least 1 T1D autoantibody
  * treatment to be started within 150 days of diagnosis
  * greater than 0.2 nmol/L of C-peptide following mixed meal tolerance test
  * No active infections
Groups:
- AG019 Cohort 1 - Low (Single) Dose/Adults; AG019 Cohort 3 - Low (Single) Dose/Adolescents: AG019 - Low Dose: Solid, orally administered capsule - 2 capsules per day for 1 day (single dose)
- AG019 Cohort 1 - Low (Repeat) Dose/Adults; AG019 Cohort 3 - Low (Repeat) Dose/Adolescents: AG019 - Low Dose: Solid, orally administered capsule - 2 capsules per day for 8 weeks (repeat dose)
- AG019 Cohort 2 - High (Single) Dose/Adults; AG019 Cohort 4 - High (Single) Dose/Adolescents: AG019 - High Dose: Solid, orally administered capsule - 6 capsules per day for 1 day (single dose)
- AG019 Cohort 2 - High (Repeat) Dose/Adults; AG019 Cohort 4 - High (Repeat) Dose/Adolescents: AG019 - High Dose: Solid, orally administered capsule - 6 capsules per day for 8 weeks (repeat dose)
- Combination Cohort 1 - Active AG019/Teplizumab - Adults; Combination Cohort 2 - Active AG019/Teplizumab - Adolescents: Teplizumab: Daily IV infusions of Teplizumab during the first 12 days of AG019 treatment. Total cumulative dose is approximately 17mg (dose calculation based on body surface area).
  AG019 - High Dose: Solid, orally administered capsule - 6 capsules per day for 8 weeks.
- Combination Cohort 1 - AG019-placebo/Teplizumab-placebo - Adults; Combination Cohort 2 - AG019-placebo/Teplizumab-placebo - Adolescents: Placebo-AG019: Formulated identically to AG019 with the active ingredient removed.
  Placebo-Teplizumab: Formulated identically to teplizumab with the active ingredient removed.
Period: Overall Study
Arm/Group | AG019 Cohort 1 - Low (Single) Dose/Adults | AG019 Cohort 1 - Low (Repeat) Dose/Adults | AG019 Cohort 2 - High (Single) Dose/Adults | AG019 Cohort 2 - High (Repeat) Dose/Adults | AG019 Cohort 3 - Low (Single) Dose/Adolescents | AG019 Cohort 3 - Low (Repeat) Dose/Adolescents | AG019 Cohort 4 - High (Single) Dose/Adolescents | AG019 Cohort 4 - High (Repeat) Dose/Adolescents | Combination Cohort 1 - Active AG019/Teplizumab - Adults | Combination Cohort 1 - AG019-placebo/Teplizumab-placebo - Adults | Combination Cohort 2 - Active AG019/Teplizumab - Adolescents | Combination Cohort 2 - AG019-placebo/Teplizumab-placebo - Adolescents
Started | 2 | 5 | 2 | 5 | 2 | 4 | 2 | 5 | 10 | 2 | 5 | 1
Completed | 2 | 5 | 2 | 4 | 2 | 4 | 2 | 4 | 10 | 2 | 4 | 0
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AG019 Cohort 1 - Low (Single) Dose/Adults | AG019 Cohort 1 - Low (Repeat) Dose/Adults | AG019 Cohort 2 - High (Single) Dose/Adults | AG019 Cohort 2 - High (Repeat) Dose/Adults | AG019 Cohort 3 - Low (Single) Dose/Adolescents | AG019 Cohort 3 - Low (Repeat) Dose/Adolescents | AG019 Cohort 4 - High (Single) Dose/Adolescents | AG019 Cohort 4 - High (Repeat) Dose/Adolescents | Combination Cohort 1 - Active AG019/Teplizumab - Adults | Combination Cohort 1 - AG019-placebo/Teplizumab-placebo - Adults | Combination Cohort 2 - Active AG019/Teplizumab - Adolescents | Combination Cohort 2 - AG019-placebo/Teplizumab-placebo - Adolescents | Total
Number analyzed (Participants) | 2 | 5 | 2 | 5 | 2 | 4 | 2 | 5 | 10 | 2 | 5 | 1 | 45
Age, Continuous [Median (Standard Deviation); unit: years] | 38.0 (5.7) | 26.0 (8.9) | 19.5 (2.1) | 22.0 (7.4) | 16.5 (0.7) | 14.0 (2.2) | 17.0 (0.0) | 14.0 (1.9) | 26.5 (6.7) | 29.0 (5.7) | 14.0 (1.1) | 12.0 (0.0) | 20.0 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2 | 2 | 2 | 0 | 3 | 4 | 1 | 3 | 1 | 20
  Male | 2 | 4 | 1 | 3 | 0 | 2 | 2 | 2 | 6 | 1 | 2 | 0 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 2 | 5 | 1 | 4 | 2 | 4 | 1 | 5 | 10 | 2 | 5 | 1 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Baseline serological cytomegalovirus positivity [Count of Participants; unit: Participants]
  Negative | 2 | 5 | 2 | 5 | 2 | 3 | 2 | 5 | 5 | 1 | 4 | 1 | 37
  Positive | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 1 | 0 | 0 | 7
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Baseline serological Epstein-Barr virus positivity [Count of Participants; unit: Participants]
  Negative | 2 | 2 | 2 | 4 | 2 | 4 | 2 | 4 | 4 | 0 | 4 | 1 | 31
  Positive | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 6 | 2 | 1 | 0 | 14
Autoantibody positivity - GAD65 [Count of Participants; unit: Participants]
  Negative | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 3
  Positive | 1 | 5 | 2 | 5 | 1 | 3 | 1 | 5 | 10 | 2 | 3 | 1 | 39
  Missing | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Autoantibody positivity - IA-2 [Count of Participants; unit: Participants]
  Negative | 1 | 2 | 1 | 1 | 0 | 2 | 0 | 2 | 5 | 1 | 1 | 0 | 16
  Positive | 0 | 2 | 1 | 4 | 1 | 2 | 0 | 2 | 3 | 1 | 4 | 1 | 21
  Missing | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 8
Autoantibody positivity - ZnT8 [Count of Participants; unit: Participants]
  Negative | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 7
  Positive | 1 | 2 | 1 | 2 | 0 | 3 | 0 | 3 | 5 | 0 | 3 | 0 | 20
  Missing | 1 | 3 | 0 | 1 | 2 | 0 | 2 | 1 | 3 | 2 | 2 | 1 | 18
Autoantibody positivity - Insulin [Count of Participants; unit: Participants]
  Negative | 1 | 2 | 1 | 2 | 0 | 1 | 1 | 2 | 5 | 1 | 3 | 0 | 19
  Positive | 0 | 3 | 1 | 3 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 1 | 13
  Missing | 1 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 5 | 0 | 1 | 0 | 13
Insulin required at baseline [Count of Participants; unit: Participants]
  Yes | 1 | 5 | 2 | 4 | 2 | 4 | 2 | 5 | 10 | 2 | 5 | 1 | 43
  No | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Baseline HbA1c [Mean (Standard Deviation); unit: percent] — Percentage of hemoglobin proteins in the blood that are glycated (i.e., the percentage of hemoglobin proteins that hold glucose). Population: this assessment was not required for single dose patients, result not available
  percent
    number analyzed (Participants) | 0 | 5 | 0 | 5 | 0 | 4 | 0 | 5 | 10 | 2 | 5 | 1 | 37
    (all) |  | 6.38 (0.56) |  | 7.00 (1.57) |  | 6.40 (0.51) |  | 6.28 (0.89) | 6.92 (1.42) | 7.35 (3.04) | 7.14 (2.43) | 8.40 | 6.86 (1.44)
Time from diagnosis to treatment [Mean (Standard Deviation); unit: days] | 84.5 (44.5) | 91.0 (38.2) | 45.5 (20.5) | 100 (42.2) | 146.0 (4.2) | 95.0 (21.3) | 113.0 (53.7) | 126.4 (19.4) | 101.0 (35.9) | 70.0 (15.6) | 122.6 (36.3) | 90.0 | 102.2 (36.1)
Baseline IDAA1c [Mean (Standard Deviation); unit: units on a scale'] — IDAA1c or insulin dose adjusted HbA1c is a calculated unit. Formula:
  IDAA1c = HbA1c (%) + 4*total daily insulin dose (IU/kg)
  IDAA1c values below or equal to 9 generally represent partial disease remission. Population: this assessment was not required for single dose patients, result not available
  units on a scale'
    number analyzed (Participants) | 0 | 5 | 0 | 5 | 0 | 4 | 0 | 5 | 10 | 2 | 5 | 1 | 37
    (all) |  | 7.385 (1.303) |  | 8.248 (2.369) |  | 9.090 (1.093) |  | 8.392 (2.470) | 8.412 (1.725) | 8.530 (4.540) | 9.605 (2.583) | 10.640 | 8.55 (2.02)
Fasting C-peptide [Mean (Standard Deviation); unit: nmol/L] — Population: this assessment was not required for single dose patients, result not available
  nmol/L
    number analyzed (Participants) | 0 | 5 | 0 | 5 | 0 | 4 | 0 | 5 | 10 | 2 | 5 | 1 | 37
    (all) |  | 0.27 (0.15) |  | 0.38 (0.19) |  | 0.33 (0.08) |  | 0.27 (0.14) | 0.18 (0.13) | 0.36 (0.22) | 0.25 (0.07) | 0.16 | 0.65 (0.46)
Peak stimulated C-peptide [Mean (Standard Deviation); unit: nmol/L] — Population: this assessment was not required for single dose patients, result not available
  nmol/L
    number analyzed (Participants) | 0 | 5 | 0 | 5 | 0 | 4 | 0 | 5 | 10 | 2 | 5 | 1 | 37
    (all) |  | 0.92 (0.35) |  | 1.26 (1.12) |  | 0.97 (0.45) |  | 0.81 (0.09) | 0.71 (0.26) | 1.10 (0.11) | 0.76 (0.25) | 0.28 | 2.08 (1.54)
Mean 2H C-peptide AUC [Mean (Standard Deviation); unit: nmol/L] — * Mixed Meal Tolerance test (MMTT)-stimulated 2-hour C-peptide area under the curve (AUC) was defined as the mean area under the C-peptide level time curve over the 2-hour period divided by the duration after an MMTT.
  * Mean 2h AUC is the AUC (expressed as nmol*min/L) divided by the number of minutes (120 min). Population: this assessment was not required for single dose patients, result not available
  nmol/L
    number analyzed (Participants) | 0 | 5 | 0 | 5 | 0 | 4 | 0 | 5 | 10 | 2 | 5 | 1 | 37
    (all) |  | 0.418 (0.257) |  | 0.500 (0.327) |  | 0.428 (0.134) |  | 0.512 (0.484) | 0.464 (0.255) | 0.396 (0.000) | 0.665 (0.160) | 0.000 (0.000) | 0.63 (0.32)
Total daily insulin use [Mean (Standard Deviation); unit: IU/kg/d] — Population: this assessment was not required for single dose patients, result not available
  IU/kg/d
    number analyzed (Participants) | 0 | 5 | 0 | 5 | 0 | 4 | 0 | 5 | 10 | 2 | 5 | 1 | 37
    (all) |  | 0.23 (0.18) |  | 0.39 (0.20) |  | 0.67 (0.27) |  | 0.53 (0.46) | 0.37 (0.14) | 0.30 (0.37) | 0.51 (0.18) | 0.56 | 0.42 (0.27)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent Adverse Events (TEAE)
Description: Treatment-emergent adverse events assessed by the investigator, review of lab reports and information provided by the participant during site visits and/or participant diary with AG019 alone or with teplizumab
Time Frame: up to 6 months
Measure: Number; unit: Events
Groups:
- Combination Cohort 1 - Active AG019/Teplizumab - Adults; Combination Cohort 2 - Active AG019/Teplizumab - Adolescents: Teplizumab: Daily IV infusions of Teplizumab during the first 12 days of AG019 treatment. Total cumulative dose is approximately 17mg (dose calculation based on body surface area).
  AG019 - High Dose: Solid, orally administered capsule - 6 capsules per day for 8 weeks (repeat dose).
Arm/Group | AG019 Cohort 1 - Low (Single) Dose/Adults | AG019 Cohort 1 - Low (Repeat) Dose/Adults | AG019 Cohort 2 - High (Single) Dose/Adults | AG019 Cohort 2 - High (Repeat) Dose/Adults | AG019 Cohort 3 - Low (Single) Dose/Adolescents | AG019 Cohort 3 - Low (Repeat) Dose/Adolescents | AG019 Cohort 4 - High (Single) Dose/Adolescents | AG019 Cohort 4 - High (Repeat) Dose/Adolescents | Combination Cohort 1 - Active AG019/Teplizumab - Adults | Combination Cohort 1 - AG019-placebo/Teplizumab-placebo - Adults | Combination Cohort 2 - Active AG019/Teplizumab - Adolescents | Combination Cohort 2 - AG019-placebo/Teplizumab-placebo - Adolescents
Number analyzed (Participants) | 2 | 5 | 2 | 5 | 2 | 4 | 2 | 5 | 10 | 2 | 5 | 1
Events | 1 | 6 | 1 | 19 | 1 | 28 | 1 | 19 | 91 | 25 | 22 | 1

2. Secondary Outcome: AG019 in Systemic Circulation
Description: The presence of live L. lactis bacteria in blood will be assessed by plating
Time Frame: Up to 3 months after initiation of the treatment
Population: This assessment was not required for single dose patients, result not available
Measure: Count of Participants; unit: Participants
Arm/Group | AG019 Cohort 1 - Low (Repeat) Dose/Adults | AG019 Cohort 2 - High (Repeat) Dose/Adults | AG019 Cohort 3 - Low (Repeat) Dose/Adolescents | AG019 Cohort 4 - High (Repeat) Dose/Adolescents | Combination Cohort 1 - Active AG019/Teplizumab - Adults | Combination Cohort 1 - AG019-placebo/Teplizumab-placebo - Adults | Combination Cohort 2 - Active AG019/Teplizumab - Adolescents | Combination Cohort 2 - AG019-placebo/Teplizumab-placebo - Adolescents
Number analyzed (Participants) | 5 | 5 | 4 | 5 | 10 | 2 | 4 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: L. Lactis-secreted hPINS or hIL-10 in Systemic Circulation
Description: The presence of L. lactis-secreted hPINS or hIL-10 in the blood will be assessed by ELISA (enzyme-linked immunosorbent assay)
Time Frame: Up to 3 months after initiation of the treatment
Population: Indication for exposure of AG019 secreted hPINS or hIL-10 protein in plasma This assessment was not required for single dose patients, result not available
Measure: Count of Participants; unit: Participants
Arm/Group | AG019 Cohort 1 - Low (Repeat) Dose/Adults | AG019 Cohort 2 - High (Repeat) Dose/Adults | AG019 Cohort 3 - Low (Repeat) Dose/Adolescents | AG019 Cohort 4 - High (Repeat) Dose/Adolescents | Combination Cohort 1 - Active AG019/Teplizumab - Adults | Combination Cohort 1 - AG019-placebo/Teplizumab-placebo - Adults | Combination Cohort 2 - Active AG019/Teplizumab - Adolescents | Combination Cohort 2 - AG019-placebo/Teplizumab-placebo - Adolescents
Number analyzed (Participants) | 5 | 5 | 4 | 5 | 10 | 2 | 4 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: AG019 in Feces
Description: The presence of L. lactis (live or dead) in feces will be assessed by Q-PCR (quantitative real-time polymerase chain reaction)
Time Frame: Up to 8 days after completion of the treatment
Population: This assessment was not required for single dose patients, result not available
Measure: Count of Participants; unit: Participants
Arm/Group | AG019 Cohort 2 - High (Repeat) Dose/Adults | AG019 Cohort 4 - High (Repeat) Dose/Adolescents | Combination Cohort 1 - Active AG019/Teplizumab - Adults | Combination Cohort 1 - AG019-placebo/Teplizumab-placebo - Adults | Combination Cohort 2 - Active AG019/Teplizumab - Adolescents | Combination Cohort 2 - AG019-placebo/Teplizumab-placebo - Adolescents
Number analyzed (Participants) | 5 | 4 | 10 | 2 | 3 | 1
Participants
  participants with AG019 in feces | 3 | 3 | 9 | 0 | 3 | 0
  participants with no AG019 in feces | 2 | 1 | 1 | 2 | 0 | 1

5. Secondary Outcome: C-peptide Area Under the Concentration-time Curve (AUC) Calculated From a 2 Hour Mixed Meal Tolerance Test (MMTT) at 12 Months
Description: MMTT-stimulated 2-hour C-peptide AUC was defined as the mean area under the C-peptide level time curve over the 2-hour period divided by the duration after a mixed-meal tolerance test.
Time Frame: up to 12 months
Measure: Mean (Standard Deviation); unit: nmol/L
Groups:
- AG019 Cohort 1 - Low (Repeat)-Dose/Adults; AG019 Cohort 3 - Low (Repeat) Dose/Adolescents: AG019 - Low Dose: Solid, orally administered capsule - 2 capsules per day for 8 weeks (repeat dose)
Arm/Group | AG019 Cohort 2 - High (Repeat) Dose/Adults | AG019 Cohort 4 - High (Repeat) Dose/Adolescents | Combination Cohort 1 - Active AG019/Teplizumab - Adults | Combination Cohort 1 - AG019-placebo/Teplizumab-placebo - Adults | Combination Cohort 2 - Active AG019/Teplizumab - Adolescents | Combination Cohort 2 - AG019-placebo/Teplizumab-placebo - Adolescents | AG019 Cohort 1 - Low (Repeat)-Dose/Adults | AG019 Cohort 3 - Low (Repeat) Dose/Adolescents
Number analyzed (Participants) | 5 | 5 | 10 | 2 | 5 | 1 | 5 | 4
nmol/L | 0.89 (0.61) | 0.57 (0.13) | 0.48 (0.19) | 0.73 (0.01) | 0.57 (0.21) | 0.25 (0) | 0.62 (0.48) | 0.78 (0.35)

6. Other Pre Specified Outcome: Incidence of Treatment Emergent Adverse Events up to 12 Months
Description: Incidence of all reported TEAE up to the 12-month follow-up visit. The TEAE are counted once within each patient on the preferred term level.
Time Frame: Up to 12 months from screening
Measure: Number; unit: events
Arm/Group | AG019 Cohort 1 - Low (Single) Dose/Adults | AG019 Cohort 1 - Low (Repeat) Dose/Adults | AG019 Cohort 2 - High (Single) Dose/Adults | AG019 Cohort 2 - High (Repeat) Dose/Adults | AG019 Cohort 3 - Low (Single) Dose/Adolescents | AG019 Cohort 3 - Low (Repeat) Dose/Adolescents | AG019 Cohort 4 - High (Single) Dose/Adolescents | AG019 Cohort 4 - High (Repeat) Dose/Adolescents | Combination Cohort 1 - Active AG019/Teplizumab - Adults | Combination Cohort 1 - AG019-placebo/Teplizumab-placebo - Adults | Combination Cohort 2 - Active AG019/Teplizumab - Adolescents | Combination Cohort 2 - AG019-placebo/Teplizumab-placebo - Adolescents
Number analyzed (Participants) | 2 | 2 | 2 | 5 | 2 | 4 | 2 | 5 | 10 | 2 | 5 | 1
events | 1 | 8 | 1 | 26 | 1 | 33 | 1 | 26 | 97 | 26 | 23 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from signature of informed consent until completion of the study (or premature withdrawal), an average of 13 months (1 month of screening plus 12 months of study participation).
Description: All adverse events are listed, regardless of treatment emergence, severity, or relationship to AG019 or teplizumab. The results of the primary endpoint (incidence of TEAE up to 6 months) are outlined in the Endpoints section.
Arm/Group | AG019 Cohort 1 - Low (Single) Dose/Adults | AG019 Cohort 1 - Low (Repeat) Dose/Adults | AG019 Cohort 2 - High (Single) Dose/Adults | AG019 Cohort 2 - High (Repeat) Dose/Adults | AG019 Cohort 3 - Low (Single) Dose/Adolescents | AG019 Cohort 3 - Low (Repeat) Dose/Adolescents | AG019 Cohort 4 - High (Single) Dose/Adolescents | AG019 Cohort 4 - High (Repeat) Dose/Adolescents | Combination Cohort 1 - Active AG019/Teplizumab - Adults | Combination Cohort 1 - AG019-placebo/Teplizumab-placebo - Adults | Combination Cohort 2 - Active AG019/Teplizumab - Adolescents | Combination Cohort 2 - AG019-placebo/Teplizumab-placebo - Adolescents
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/5 | 0/2 | 0/5 | 0/2 | 0/4 | 0/2 | 0/5 | 0/10 | 0/2 | 0/5 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/5 | 0/2 | 0/5 | 0/2 | 0/4 | 0/2 | 0/5 | 0/10 | 0/2 | 0/5 | 0/1
Other Adverse Events (participants affected / at risk) | 1/2 | 3/5 | 1/2 | 2/5 | 1/2 | 2/4 | 1/2 | 2/5 | 5/10 | 2/2 | 2/5 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AG019 Cohort 1 - Low (Single) Dose/Adults (N=2) | AG019 Cohort 1 - Low (Repeat) Dose/Adults (N=5) | AG019 Cohort 2 - High (Single) Dose/Adults (N=2) | AG019 Cohort 2 - High (Repeat) Dose/Adults (N=5) | AG019 Cohort 3 - Low (Single) Dose/Adolescents (N=2) | AG019 Cohort 3 - Low (Repeat) Dose/Adolescents (N=4) | AG019 Cohort 4 - High (Single) Dose/Adolescents (N=2) | AG019 Cohort 4 - High (Repeat) Dose/Adolescents (N=5) | Combination Cohort 1 - Active AG019/Teplizumab - Adults (N=10) | Combination Cohort 1 - AG019-placebo/Teplizumab-placebo - Adults (N=2) | Combination Cohort 2 - Active AG019/Teplizumab - Adolescents (N=5) | Combination Cohort 2 - AG019-placebo/Teplizumab-placebo - Adolescents (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 1 (1) | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Erythropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 (1) | 0 | 2 (3) | 0 | 2 (2) | 2 (3) | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0 | 1 (1) | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (6) | 0 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 (1) | 0 | 1 (3) | 0 | 0 | 3 (5) | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Coeliac disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (2) | 0 | 1 (1) | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 2 (4) | 0 | 1 (1) | 0 | 0 | 4 (4) | 1 (1) | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Glossitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 0 | 1 (1) | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Tongue dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (3) | 4 (12) | 0 | 2 (2) | 0
Administration site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Catheter site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Catheter site related reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 2 (2) | 1 (3) | 1 (1) | 0
Influenza like illness (General disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site irritation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 2 (2) | 1 (1) | 1 (2) | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Selective IgA immunodeficiency (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Body tinea (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Medical device site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 (3) | 0 | 1 (2) | 0 | 0 | 0 | 0 | 3 (3) | 1 (1) | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 3 (4) | 0 | 1 (2) | 0 | 2 (2) | 0 | 2 (4) | 1 (1) | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 (3) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Joint Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 (2) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 1 (1) | 0
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (2) | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (2) | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body Temperature decreased (Investigations) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Epstein-Barr virus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 2 (4) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (3) | 0 | 2 (2) | 0
Monocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Protein total increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 (2) | 0 | 1 (1) | 0 | 1 (1) | 0 | 0 | 1 (1) | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 (3) | 1 (8) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (0) | 1 (1) | 1 (1) | 0 | 0
Growing pains (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (2) | 0 | 0 | 0 | 0
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (5) | 0 | 2 (2) | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 (2) | 0 | 0 | 1 (2) | 0 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (2) | 5 (7) | 2 (11) | 1 (3) | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 1 (1) | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 0 | 1 (1) | 1 (1)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Scrotal irritation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (2) | 1 (1) | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 2 (2) | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 2 (6) | 1 (1) | 0 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 (5) | 0 | 1 (1) | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (2) | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
haemoglobin increased (Investigations) | 0 | 0 | 0 | 1 (2) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Confidentiality and consulting agreements restrict the dissemination of confidential information, but PIs are not restricted to act as a consultant for other companies.

DOCUMENTS (2):
  • Study Protocol (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/07/NCT03751007/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT03751007/SAP_001.pdf